CLINICAL TRIAL: NCT03187327
Title: Feasibility of Opportunistic Salpingectomy at the Time of Vaginal Hysterectomy for Benign Pathology and Evaluation of Occult Tubal Lesions Prevalence: Preliminary Study
Brief Title: Feasibility of Opportunistic Salpingectomy at the Time of Vaginal Hysterectomy for Benign Pathology
Acronym: FPS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0352
Record Dates: First submitted 2017-06-13; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Salpingectomy; Hysterectomy
Keywords: prophylactic salpingectomy; vaginal hysterectomy; p53 expression; ovarian cancers
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this prospective study, patients who underwent vaginal hysterectomy with salpingectomy or salpingo-oophorectomy were included. The objective of this study is to assess the feasibility of prophylactic salpingectomy during vaginal hysterectomy for benign pathology and the prevalence of occult tubal lesions. The hypothesis is that prophylactic salpingectomy during vaginal hysterectomy for benign pathology present a low failure rate and it makes it possible to avoid the appearance of a certain number of ovarian cancers. The prevalence of bilateral salpingectomy with or without ovariectomy and the prevalence of histopathological and immunohistochemical (p53 expression) abnormalities were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent vaginal hysterectomy for benign pathology with salpingectomy or salpingo-oophorectomy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent vaginal hysterectomy with salpingectomy or salpingo-oophorectomy
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Success rate of the surgical technique | Day 0
  prevalence of bilateral salpingectomy with or without ovariectomy

CONTACTS AND LOCATIONS:
Overall Officials: Gautier CHENE, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Femme Mère Enfant, Bron, France

IPD SHARING:
Plan to Share IPD: No